CLINICAL TRIAL: NCT03724253
Title: Phase II Study of Preliminary Diagnostic Performance of [68Ga]-NeoBOMB1 in Adult Patients With Malignancies Known to Overexpress Gastrin Releasing Peptide Receptor (GRPR)
Brief Title: [68Ga]-NeoBOMB1 Imaging in Patients With Malignancies Known to Overexpress Gastrin Releasing Peptide Receptor (GRPR)
Acronym: NeoFIND
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Recruitment was stopped before the target sample size was achieved.
Sponsor: Advanced Accelerator Applications (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: A005D-E01-201; 2017-003432-37 (EudraCT Number); CAAA503A12201 (Other: Novartis)
Record Dates: First submitted 2018-10-21; First posted 2018-10-30 (Actual); Results first posted 2020-10-23 (Actual); Last update posted 2020-10-23 (Actual); Status verified 2020-10

CONDITIONS: Breast Cancer; Prostate Cancer; Colorectal Cancer; Non Small Cell Lung Cancer; Small Cell Lung Cancer
Keywords: [68Ga]-NeoBOMB1
MeSH Terms: conditions — Breast Neoplasms; Prostatic Neoplasms; Colorectal Neoplasms; Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma

STUDY DESIGN:
Intervention Model Description: The study design included a dosimetry and non-dosimetry groups and with the following tumor types:
  * Breast Cancer: dosimetry and non-dosimetry groups
  * Prostate Cancer: dosimetry and non-dosimetry groups
  * Colorectal cancer: non-dosimetry group
  * Non-Small Cell Lung Cancer (NSCLC): non-dosimetry group
  * Small-Cell Lung Cancer (SCLC): non-dosimetry group All data presentations were to be presented primarily by the overall population but were also to be repeated split by tumor type where relevant. Some presentations were also to be repeated split by whether or not the patient was found to have tumors bearing GRPR expression according to cytology and/or histopathology findings.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase II dosimetry group (Experimental): All eligible participants were to receive recommended dose of [68Ga]-NeoBOMB1 of 3 Mega Becquerel (MBq)/Kg (+/- 10%) [but not more than 250 and not less than 150 MBq. The maximum peptide mass administered was 50 microgram (µg)].
  Interventions: Drug: [68Ga]-NeoBOMB1
- Phase II non-dosimetry group (Experimental): All eligible participants were to receive recommended dose of [68Ga]-NeoBOMB1 of 3 Mega Becquerel (MBq)/Kg (+/- 10%) [but not more than 250 and not less than 150 MBq. The maximum peptide mass administered was 50 microgram (µg)].
  Interventions: Drug: [68Ga]-NeoBOMB1

INTERVENTIONS:
Drug: [68Ga]-NeoBOMB1 — [68Ga]-radiolabeled bombesin peptide targeting Gastrin Releasing Peptide Receptors

SUMMARY:
This was a Phase II, multi-center, open label, single dose study in patients with tumor types known to overexpress Gastrin-Releasing Peptide Receptor (GRPR), including breast, prostate, colorectal, Non-Small Cell Lung Cancer (NSCLC) and Small-Cell Lung Cancer (SCLC).

DETAILED DESCRIPTION:
A total of 50 subjects were planned for the study (10 subjects for the dosimetry group and 40 subjects for the non dosimetry group). In total, 22 subjects were screened for eligibility and 19 subjects were enrolled (2 subjects in the dosimetry group and 17 subjects in the non dosimetry group).

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be at least 18 years of age
* Subjects must have signed and dated an informed consent prior to any study-specific procedures
* Subjects with histologically-confirmed tumor for whom a recent biopsy (not older than 6-months old) has been performed.
* Dosimetry group: luminal breast cancer, adenocarcinoma of the prostate
* Non-dosimetry group: luminal breast cancer, adenocarcinoma of the prostate, small cell lung cancer, non-small cell lung cancer, colorectal carcinoma
* At least one malignant lesion detected via functional or morphological imaging (PET combined to appropriate tracer according to tumor type, CT, MRI) within 3 months prior to [68Ga]-NeoBOMB1 administration
* The Eastern Cooperative Oncology (ECOG) performance status 0-2.
* Subjects must agree to use highly effective methods of contraception (female partners of male participants should use highly effective methods of contraception) during the trial.

Exclusion Criteria:

* renal insufficiency or an eGFR <50 ml/min/1.73m2
* hematological toxicity grade > 2 (Toxicity Grading Scale in vaccine clinical trials)
* participation in any other investigational trial within 30 days of study entry
* subjects with positive pregnancy test (urine dipstick), and/or currently breast-feeding
* concurrent severe illness or clinically relevant trauma within 2 weeks before the administration of the investigational product that might preclude study completion or interfere with study results
* concurrent bladder outflow obstruction or unmanageable urinary incontinence
* known or expected hypersensitivity to [68Ga]-NeoBOMB1 or any excipient present in [68Ga]-NeoBOMB1
* any condition that precludes raised arms position
* prior administration of a radiopharmaceutical within a period corresponding to 8 half-lives of the radionuclide
* history of somatic or psychiatric disease/condition that may interfere with the objectives and assessments of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2018-07-03 (Actual); Primary Completion 2019-06-20 (Actual); Study Completion 2019-07-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (3):
- Medical University Innsbruck Department of Nuclear Medicine, Innsbruck, Austria
- France (2):
  - University of Grenoble - Hopital Michallon, Service de Medicine Nucleaire, La Tronche
  - University of Bordeaux, Unite TEP RECHERCHE - Hopital Xavier Arnozan, Pessac

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 3 centers in 2 countries: Austria (1) and France (2).
Pre-assignment Details: A total of 50 subjects were planned for the study (10 subjects for the dosimetry group and 40 subjects for the non dosimetry group). In total, 22 subjects were screened for eligibility and 19 subjects were enrolled (2 subjects in the dosimetry group and 17 subjects in the non dosimetry group).
Groups:
- Breast; Prostate; Colorectal; Non-Small Cell Lung Cancer (NSCLC); Small-Cell Lung Cancer (SCLC): All eligible participants were to receive recommended dose of [68Ga]-NeoBOMB1 of 3 Mega Becquerel (MBq)/Kg (+/- 10%) [but not more than 250 and not less than 150 MBq. The maximum peptide mass administered was 50 microgram (µg)].
Period: Overall Study
Arm/Group | Breast | Prostate | Colorectal | Non-Small Cell Lung Cancer (NSCLC) | Small-Cell Lung Cancer (SCLC)
Started (Full Analysis Set (FAS) = all subjects who enter the study and receive the [68Ga]-NeoBOMB1 dose) | 5 | 5 | 5 | 3 | 1
Completed | 5 | 5 | 5 | 3 | 1
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) = all subjects who enter the study and receive the [68Ga]-NeoBOMB1 dose.
Groups:
- Total: Total of all reporting groups
Arm/Group | Breast | Prostate | Colorectal | Non-Small Cell Lung Cancer (NSCLC) | Small-Cell Lung Cancer (SCLC) | Total
Number analyzed (Participants) | 5 | 5 | 5 | 3 | 1 | 19
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.8 (7.60) | 65.4 (6.31) | 64.2 (13.68) | 64.7 (3.21) | 54.0 (NA) — Only one participant analyzed | 63.4 (8.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 0 | 1 | 1 | 1 | 8
  Male | 0 | 5 | 4 | 2 | 0 | 11
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 0 | 2 | 3 | 2 | 1 | 8
  Not Collected | 5 | 3 | 2 | 1 | 0 | 11
Baseline Weight [Mean (Standard Deviation); unit: kilogram (kg)] — Baseline is defined as the last measurement prior to Investigational Medicinal Product (IMP) administration.
  kilogram (kg) | 70.6 (10.53) | 85.2 (7.46) | 72.6 (8.63) | 72.1 (23.38) | 62.8 (NA) — Only one participant analyzed | 74.8 (12.64)
Baseline Height [Mean (Standard Deviation); unit: centimeter (cm)] — Baseline is defined as the last measurement prior to Investigational Medicinal Product (IMP) administration.
  centimeter (cm) | 165.6 (3.21) | 175.4 (5.94) | 170.4 (6.23) | 165.7 (3.51) | 168.0 (NA) — Only one participant analyzed | 169.6 (10.7)
Baseline Body Mass Index [Mean (Standard Deviation); unit: kilogram per square metre (kg/m^2)] — Baseline is defined as the last measurement prior to Investigational Medicinal Product (IMP) administration.
  kilogram per square metre (kg/m^2) | 25.84 (4.563) | 27.79 (3.202) | 24.90 (1.514) | 26.04 (7.552) | 22.25 (NA) — Only one participant analyzed | 25.95 (3.970)
Diagnostic Stage [Count of Participants; unit: Participants] — The overall diagnostic stage uses the stage at screening visit and the Tumour, Node, Metastasis (TNM) staging uses the latest available stage. Stage III indicates a locally advanced cancer that is likely to grow and spread; stage IIIA = the cancer has spread into nearby tissues; stage IIIC = the cancer cells across the tumor are poorly differentiated, meaning they look very different from healthy cells. Stage IV means that the cancer has spread to distant parts of the body and may be called advanced or metastatic cancer.
  Participants
    IIIA | 0 | 1 | 0 | 1 | 0 | 2
    IIIC | 0 | 0 | 0 | 1 | 0 | 1
    IV | 5 | 4 | 5 | 1 | 1 | 16
Time from Initial Diagnosis of Primary Disease [Mean (Standard Deviation); unit: Months] — Time from initial diagnosis (months) is calculated as (date of IMP administration - date of initial diagnosis + 1)/30.4375.
  Months | 117.3 (64.61) | 50.5 (74.48) | 24.3 (25.40) | 1.6 (1.46) | 1.1 (NA) — Only one participant analyzed | 50.9 (65.32)

OUTCOME MEASURES:

1. Primary Outcome: Number of Lesions Detected by [68Ga]-NeoBOMB1
Description: The preliminary targeting properties of [68Ga]-NeoBOMB1 were to be assessed by summarizing the number of lesions identified by Positron Emission Tomography (PET) overall and split by GRPR positive and negative patients, as well as by tumor type. Only descriptive analysis performed.
Time Frame: [68Ga]-NeoBOMB1 PET imaging acquired at Day 1
Population: Full Analysis Set (FAS). The results of the biopsied samples for all patients were positive for GRPR and thus the presentation of results according to GRPR expression were no longer suitable.
Measure: Mean (Standard Deviation); unit: Lesion
Arm/Group | Breast | Prostate | Colorectal | Non-Small Cell Lung Cancer (NSCLC) | Small-Cell Lung Cancer (SCLC)
Number analyzed (Participants) | 5 | 5 | 5 | 3 | 1
Lesion | 17.0 (15.57) | 2.2 (1.64) | 6.0 (4.58) | 3.3 (2.31) | 1.0 (NA) — Only one participant analyzed

2. Primary Outcome: Number of Participants With Lesions Detected by [68Ga]-NeoBOMB1 Per Location
Description: The preliminary targeting properties of [68Ga]-NeoBOMB1 were to be assessed by summarizing the location of lesions identified by PET overall and split by GRPR positive and negative patients, as well as by tumor type. Only descriptive analysis performed.
Time Frame: [68Ga]-NeoBOMB1 PET imaging acquired at Day 1
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Breast | Prostate | Colorectal | Non-Small Cell Lung Cancer (NSCLC) | Small-Cell Lung Cancer (SCLC)
Number analyzed (Participants) | 5 | 5 | 3 | 3 | 1
Participants
  Overall | 5 | 5 | 3 | 3 | 1
  Nodal | 2 | 1 | 2 | 3 | 0
  Skeletal | 4 | 2 | 0 | 0 | 0
  Skin/Superficial | 2 | 0 | 0 | 0 | 0
  Soft Tissue/Visceral | 4 | 4 | 2 | 3 | 1

3. Primary Outcome: Non-Dosimetry Group: Standard Uptake Value (SUV) Mean by Timepoint and Lesion Location
Description: Targeting properties of [68Ga]-NeoBOMB1 were to be evaluated by semi-quantitatively assessing radiotracer uptake at lesion level, identified via PET Imaging. The SUVmean and SUVmax (g/mL) of each lesion were to be calculated and reported by lesion location with summary statistics at all imaging time points. SUV was to be calculated overall and split by GRPR positive and negative patients, as well as by tumor type. Only descriptive analysis performed.
Time Frame: [68Ga]-NeoBOMB1 PET imaging acquired at Day 1 (0.05 (only applicable for the Prostate Group), 1.50 and 2.50 hours)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Standard Uptake Value (SUV)
Arm/Group | Breast | Prostate | Colorectal | Non-Small Cell Lung Cancer (NSCLC) | Small-Cell Lung Cancer (SCLC)
Number analyzed (Participants) | 5 | 5 | 5 | 3 | 1
Standard Uptake Value (SUV)
  SUV mean:Overall (0.05 hours): number analyzed (Participants) | 0 | 5 | 0 | 0 | 0
  SUV mean:Overall (0.05 hours) |  | 1.634 (0.8221) |  |  |
  SUV mean:Nodal (0.05 hours): number analyzed (Participants) | 0 | 1 | 0 | 0 | 0
  SUV mean:Nodal (0.05 hours) |  | 0.630 (NA) — Only one participant analyzed |  |  |
  SUV mean:Skeletal (0.05 hours): number analyzed (Participants) | 0 | 1 | 0 | 0 | 0
  SUV mean:Skeletal (0.05 hours) |  | 1.890 (NA) — Only one participant analyzed |  |  |
  SUV mean:Skin/Superficial (0.05 hours): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  SUV mean:Soft Tissue/Visceral (0.05 hours): number analyzed (Participants) | 0 | 4 | 0 | 0 | 0
  SUV mean:Soft Tissue/Visceral (0.05 hours) |  | 1.558 (0.9517) |  |  |
  SUV mean:Overall (1.50 hours): number analyzed (Participants) | 3 | 5 | 5 | 3 | 1
  SUV mean:Overall (1.50 hours) | 6.833 (5.0645) | 11.638 (15.9172) | 2.582 (0.8142) | 1.560 (0.4468) | 1.250 (NA) — Only one participant analyzed
  SUV mean:Nodal (1.50 hours): number analyzed (Participants) | 2 | 2 | 2 | 3 | 1
  SUV mean:Nodal (1.50 hours) | 4.720 (5.4447) | 1.080 (0.2263) | 1.700 (0.3960) | 1.560 (0.4468) | 1.250 (NA) — Only one participant analyzed
  SUV mean:Skeletal (1.50 hours): number analyzed (Participants) | 2 | 2 | 0 | 0 | 0
  SUV mean:Skeletal (1.50 hours) | 3.670 (4.0164) | 1.470 (0.7778) |  |  |
  SUV mean:Skin/Superficial (1.50 hours): number analyzed (Participants) | 1 | 0 | 1 | 0 | 0
  SUV mean:Skin/Superficial (1.50 hours) | 4.370 (NA) — Only one participant analyzed |  | 0.560 (NA) — Only one participant analyzed |  |
  SUV mean:Soft Tissue/Visceral (1.50 hours): number analyzed (Participants) | 3 | 4 | 5 | 3 | 1
  SUV mean:Soft Tissue/Visceral (1.50 hours) | 6.833 (5.0645) | 14.043 (17.2993) | 2.582 (0.8142) | 1.427 (0.4274) | 1.150 (NA) — Only one participant analyzed
  SUV mean:Overall (2.50 hours): number analyzed (Participants) | 3 | 5 | 5 | 3 | 1
  SUV mean:Overall (2.50 hours) | 6.903 (5.4174) | 9.088 (10.7319) | 2.258 (0.9105) | 1.273 (0.2386) | 0.850 (NA) — Only one participant analyzed
  SUV mean:Nodal (2.50 hours): number analyzed (Participants) | 2 | 2 | 2 | 3 | 1
  SUV mean:Nodal (2.50 hours) | 4.900 (6.0528) | 0.800 (0.2687) | 2.715 (1.5344) | 1.273 (0.2386) | 0.850 (NA) — Only one participant analyzed
  SUV mean:Skeletal (2.50 hours): number analyzed (Participants) | 2 | 2 | 0 | 0 | 0
  SUV mean:Skeletal (2.50 hours) | 3.685 (4.4336) | 1.455 (0.8415) |  |  |
  SUV mean:Skin/Superficial (2.50 hours): number analyzed (Participants) | 1 | 0 | 1 | 0 | 0
  SUV mean:Skin/Superficial (2.50 hours) | 4.360 (NA) — Only one participant analyzed |  | 0.450 (NA) — Only one participant analyzed |  |
  SUV mean:Soft Tissue/Visceral (2.50 hours): number analyzed (Participants) | 3 | 4 | 5 | 3 | 1
  SUV mean:Soft Tissue/Visceral (2.50 hours) | 6.903 (5.4174) | 10.848 (11.5294) | 2.060 (0.5115) | 1.193 (0.3250) | 0.710 (NA) — Only one participant analyzed

4. Primary Outcome: Non-Dosimetry Group: Standard Uptake Value (SUV) Max by Timepoint and Lesion Location
Description: as for outcome 3
Time Frame: [68Ga]-NeoBOMB1 PET imaging acquired at Day 1 (0.05 (only applicable for the Prostate Group), 1.50 and 2.50 hours)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Standard Uptake Value (SUV)
Arm/Group | Breast | Prostate | Colorectal | Non-Small Cell Lung Cancer (NSCLC) | Small-Cell Lung Cancer (SCLC)
Number analyzed (Participants) | 5 | 5 | 5 | 3 | 1
Standard Uptake Value (SUV)
  SUV max:Overall (0.05 hours): number analyzed (Participants) | 0 | 5 | 0 | 0 | 0
  SUV max:Overall (0.05 hours) |  | 2.166 (1.1164) |  |  |
  SUV max:Nodal (0.05 hours): number analyzed (Participants) | 0 | 1 | 0 | 0 | 0
  SUV max:Nodal (0.05 hours) |  | 0.880 (NA) — Only one participant analyzed |  |  |
  SUV max:Skeletal (0.05 hours): number analyzed (Participants) | 0 | 1 | 0 | 0 | 0
  SUV max:Skeletal (0.05 hours) |  | 2.480 (NA) — Only one participant analyzed |  |  |
  SUV max:Skin/Superficial (0.05 hours): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  SUV max:Soft Tissue/Visceral (0.05 hours): number analyzed (Participants) | 0 | 4 | 0 | 0 | 0
  SUV max:Soft Tissue/Visceral (0.05 hours) |  | 2.088 (1.2731) |  |  |
  SUV max:Overall (1.50 hours): number analyzed (Participants) | 3 | 5 | 5 | 3 | 1
  SUV max:Overall (1.50 hours) | 19.040 (17.5106) | 17.326 (24.2165) | 3.570 (0.7504) | 2.097 (0.6863) | 1.810 (NA) — Only one participant analyzed
  SUV max:Nodal (1.50 hours): number analyzed (Participants) | 2 | 2 | 2 | 3 | 1
  SUV max:Nodal (1.50 hours) | 9.070 (11.3986) | 1.505 (0.4313) | 2.090 (0.5233) | 1.917 (0.7139) | 1.450 (NA) — Only one participant analyzed
  SUV max:Skeletal (1.50 hours): number analyzed (Participants) | 2 | 2 | 0 | 0 | 0
  SUV max:Skeletal (1.50 hours) | 10.325 (13.0461) | 2.135 (0.9687) |  |  |
  SUV max:Skin/Superficial (1.50 hours): number analyzed (Participants) | 1 | 0 | 1 | 0 | 0
  SUV max:Skin/Superficial (1.50 hours) | 7.400 (NA) — Only one participant analyzed |  | 0.750 (NA) — Only one participant analyzed |  |
  SUV max:Soft Tissue/Visceral (1.50 hours): number analyzed (Participants) | 3 | 4 | 5 | 3 | 1
  SUV max:Soft Tissue/Visceral (1.50 hours) | 18.580 (17.5086) | 20.953 (26.3485) | 3.570 (0.7504) | 2.097 (0.6863) | 1.810 (NA) — Only one participant analyzed
  SUV max:Overall (2.50 hours): number analyzed (Participants) | 3 | 5 | 5 | 3 | 1
  SUV max:Overall (2.50 hours) | 23.120 (19.7908) | 14.544 (18.4921) | 2.890 (0.5866) | 2.050 (0.8314) | 1.390 (NA) — Only one participant analyzed
  SUV max:Nodal (2.50 hours): number analyzed (Participants) | 2 | 2 | 2 | 3 | 1
  SUV max:Nodal (2.50 hours) | 10.440 (13.8169) | 1.305 (0.3323) | 2.870 (1.3859) | 1.783 (0.6676) | 1.180 (NA) — Only one participant analyzed
  SUV max:Skeletal (2.50 hours): number analyzed (Participants) | 2 | 2 | 0 | 0 | 0
  SUV max:Skeletal (2.50 hours) | 15.475 (20.9091) | 2.115 (1.0677) |  |  |
  SUV max:Skin/Superficial (2.50 hours): number analyzed (Participants) | 1 | 0 | 1 | 0 | 0
  SUV max:Skin/Superficial (2.50 hours) | 7.950 (NA) — Only one participant analyzed |  | 0.600 (NA) — Only one participant analyzed |  |
  SUV max:Soft Tissue/Visceral (2.50 hours): number analyzed (Participants) | 3 | 4 | 5 | 3 | 1
  SUV max:Soft Tissue/Visceral (2.50 hours) | 22.140 (19.3278) | 17.463 (19.9790) | 2.890 (0.5866) | 2.000 (0.8982) | 1.390 (NA) — Only one participant analyzed

5. Primary Outcome: Dosimetry Group: Standard Uptake Value (SUV) Mean by Timepoint and Lesion Location
Description: as for outcome 3
Time Frame: [68Ga]-NeoBOMB1 PET imaging acquired at Day 1 (0.15, 1.00, 2.00 and 4.00 hours)
Population: Full Analysis Set (FAS). Dosimetry group targeted participants with Breast Cancer and Prostate Cancer, but only 2 participants from Breast Cancer arm enrolled in the Dosimetry Group. The results of the biopsied samples for all patients were positive for GRPR and thus the presentation of results according to GRPR expression were no longer suitable.
Measure: Mean (Standard Deviation); unit: Standard Uptake Value (SUV)
Arm/Group | Breast
Number analyzed (Participants) | 2
Standard Uptake Value (SUV)
  SUV mean:Overall (0.15 hours) | 5.615 (5.1265)
  SUV mean:Nodal (0.15 hours) | 2.565 (1.0394)
  SUV mean:Skeletal (0.15 hours) | 2.140 (0.2121)
  SUV mean:Skin/Superficial (0.15 hours): number analyzed (Participants) | 1
  SUV mean:Skin/Superficial (0.15 hours) | 1.250 (NA) — Only one participant analyzed
  SUV mean:Soft Tissue/Visceral (0.15 hours): number analyzed (Participants) | 1
  SUV mean:Soft Tissue/Visceral (0.15 hours) | 9.240 (NA) — Only one participant analyzed
  SUV mean:Overall (1.00 hours) | 4.840 (5.1336)
  SUV mean:Nodal (1.00 hours) | 2.035 (1.1667)
  SUV mean:Skeletal (1.00 hours) | 1.935 (1.2233)
  SUV mean:Skin/Superficial (1.00 hours): number analyzed (Participants) | 1
  SUV mean:Skin/Superficial (1.00 hours) | 1.520 (NA) — Only one participant analyzed
  SUV mean:Soft Tissue/Visceral (1.00 hours): number analyzed (Participants) | 1
  SUV mean:Soft Tissue/Visceral (1.00 hours) | 8.470 (NA) — Only one participant analyzed
  SUV mean:Overall ( 2.00 hours) | 4.935 (5.4659)
  SUV mean:Nodal ( 2.00 hours) | 1.865 (1.1667)
  SUV mean:Skeletal ( 2.00 hours) | 1.635 (0.7990)
  SUV mean:Skin/Superficial ( 2.00 hours): number analyzed (Participants) | 1
  SUV mean:Skin/Superficial ( 2.00 hours) | 1.650 (NA) — Only one participant analyzed
  SUV mean:Soft Tissue/Visceral ( 2.00 hours): number analyzed (Participants) | 1
  SUV mean:Soft Tissue/Visceral ( 2.00 hours) | 8.800 (NA) — Only one participant analyzed
  SUV mean:Overall ( 4.00 hours) | 5.105 (5.7064)
  SUV mean:Nodal ( 4.00 hours) | 1.475 (1.0819)
  SUV mean:Skeletal ( 4.00 hours) | 1.930 (1.2162)
  SUV mean:Skin/Superficial ( 4.00 hours): number analyzed (Participants) | 1
  SUV mean:Skin/Superficial ( 4.00 hours) | 1.100 (NA) — Only one participant analyzed
  SUV mean:Soft Tissue/Visceral ( 4.00 hours): number analyzed (Participants) | 1
  SUV mean:Soft Tissue/Visceral ( 4.00 hours) | 9.140 (NA) — Only one participant analyzed

6. Primary Outcome: Dosimetry Group: Standard Uptake Value (SUV) Max by Timepoint and Lesion Location
Description: as for outcome 3
Time Frame: [68Ga]-NeoBOMB1 PET imaging acquired at Day 1 (0.15, 1.00, 2.00 and 4.00 hours)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Standard Uptake Value (SUV)
Arm/Group | Breast
Number analyzed (Participants) | 2
Standard Uptake Value (SUV)
  SUV max:Overall( 0.15 hours) | 7.575 (6.7104)
  SUV max:Nodal (0.15 hours) | 3.405 (0.8132)
  SUV max:Skeletal (0.15 hours) | 2.740 (0.3111)
  SUV max:Skin/Superficial (0.15 hours): number analyzed (Participants) | 1
  SUV max:Skin/Superficial (0.15 hours) | 1.450 (NA) — Only one participant analyzed
  SUV max:Soft Tissue/Visceral (0.15 hours): number analyzed (Participants) | 1
  SUV max:Soft Tissue/Visceral (0.15 hours) | 12.320 (NA) — Only one participant analyzed
  SUV max:Overall (1.00 hours) | 11.550 (13.7603)
  SUV max:Nodal (1.00 hours) | 2.660 (1.1879)
  SUV max:Skeletal (1.00 hours) | 2.595 (1.5203)
  SUV max:Skin/Superficial (1.00 hours): number analyzed (Participants) | 1
  SUV max:Skin/Superficial (1.00 hours) | 1.750 (NA) — Only one participant analyzed
  SUV max:Soft Tissue/Visceral (1.00 hours): number analyzed (Participants) | 1
  SUV max:Soft Tissue/Visceral (1.00 hours) | 21.280 (NA) — Only one participant analyzed
  SUV max:Overall ( 2.00 hours) | 13.680 (17.1827)
  SUV max:Nodal ( 2.00 hours) | 2.625 (1.5486)
  SUV max:Skeletal ( 2.00 hours) | 2.445 (1.3081)
  SUV max:Skin/Superficial ( 2.00 hours): number analyzed (Participants) | 1
  SUV max:Skin/Superficial ( 2.00 hours) | 2.080 (NA) — Only one participant analyzed
  SUV max:Soft Tissue/Visceral ( 2.00 hours): number analyzed (Participants) | 1
  SUV max:Soft Tissue/Visceral ( 2.00 hours) | 25.830 (NA) — Only one participant analyzed
  SUV max:Overall ( 4.00 hours) | 13.950 (17.5787)
  SUV max:Nodal ( 4.00 hours) | 2.050 (1.3011)
  SUV max:Skeletal ( 4.00 hours) | 3.205 (2.3829)
  SUV max:Skin/Superficial ( 4.00 hours): number analyzed (Participants) | 1
  SUV max:Skin/Superficial ( 4.00 hours) | 1.640 (NA) — Only one participant analyzed
  SUV max:Soft Tissue/Visceral ( 4.00 hours): number analyzed (Participants) | 1
  SUV max:Soft Tissue/Visceral ( 4.00 hours) | 26.380 (NA) — Only one participant analyzed

7. Primary Outcome: Dosimetry Group: Evaluation of Percentage of Injected Dose Reaching the Target (TACs) in Tumors
Description: For patients included in the dosimetry group, the percentage of injected dose per gram of tissue (%ID/g) reaching tumor lesions was to be calculated using the acquired PET images at each time point. The resulting TACs were to be summarized descriptively.
Time Frame: [68Ga]-NeoBOMB1 PET imaging acquired at Day 1 (0.15, 1.00, 2.00 and 4.00 hours)
Population: Full Analysis Set (FAS). Dosimetry group targeted participants with Breast Cancer and Prostate Cancer, but only 2 participants from Breast Cancer arm enrolled in the Dosimetry Group. Due to the sample size in the dosimetry group (2 patients), summary statistics were not performed.
Measure: Number; unit: %ID/g
Arm/Group | Breast
Number analyzed (Participants) | 2
%ID/g
  Participant 1: 15 min post-dose (T1 Chest): number analyzed (Participants) | 1
  Participant 1: 15 min post-dose (T1 Chest) | 0.00347
  Participant 1: 15 min post-dose (T2 Left rib): number analyzed (Participants) | 1
  Participant 1: 15 min post-dose (T2 Left rib) | 0.00384
  Participant 1: 15 min post-dose (T3 Spine): number analyzed (Participants) | 1
  Participant 1: 15 min post-dose (T3 Spine) | 0.00469
  Participant 1: 1 hour post-dose (T1 Chest): number analyzed (Participants) | 1
  Participant 1: 1 hour post-dose (T1 Chest) | 0.00218
  Participant 1: 1 hour post-dose (T2 Left rib): number analyzed (Participants) | 1
  Participant 1: 1 hour post-dose (T2 Left rib) | 0.00251
  Participant 1: 1 hour post-dose (T3 Spine): number analyzed (Participants) | 1
  Participant 1: 1 hour post-dose (T3 Spine) | 0.00225
  Participant 1: 2 hours post-dose (T1 Chest): number analyzed (Participants) | 1
  Participant 1: 2 hours post-dose (T1 Chest) | 0.00149
  Participant 1: 2 hours post-dose (T2 Left rib): number analyzed (Participants) | 1
  Participant 1: 2 hours post-dose (T2 Left rib) | 0.00173
  Participant 1: 2 hours post-dose (T3 Spine): number analyzed (Participants) | 1
  Participant 1: 2 hours post-dose (T3 Spine) | 0.00185
  Participant 1: 4 hours post-dose (T1 Chest): number analyzed (Participants) | 1
  Participant 1: 4 hours post-dose (T1 Chest) | 0.00129
  Participant 1: 4 hours post-dose (T2 Left rib): number analyzed (Participants) | 1
  Participant 1: 4 hours post-dose (T2 Left rib) | 0.00167
  Participant 1: 4 hours post-dose (T3 Spine): number analyzed (Participants) | 1
  Participant 1: 4 hours post-dose (T3 Spine) | 0.00195
  Participant 2: 15 min post-dose (T1 lungL): number analyzed (Participants) | 1
  Participant 2: 15 min post-dose (T1 lungL) | 0.00367
  Participant 2: 15 min post-dose (T2 lungR): number analyzed (Participants) | 1
  Participant 2: 15 min post-dose (T2 lungR) | 0.00466
  Participant 2: 15 min post-dose (T3 liverL): number analyzed (Participants) | 1
  Participant 2: 15 min post-dose (T3 liverL) | 0.01353
  Participant 2: 15 min post-dose (T4 liverR1): number analyzed (Participants) | 1
  Participant 2: 15 min post-dose (T4 liverR1) | 0.01304
  Participant 2: 15 min post-dose (T5 liverR2): number analyzed (Participants) | 1
  Participant 2: 15 min post-dose (T5 liverR2) | 0.01504
  Participant 2: 15 min post-dose (T6 sacrumL): number analyzed (Participants) | 1
  Participant 2: 15 min post-dose (T6 sacrumL) | 0.00315
  Participant 2: 15 min post-dose (T7 liverP): number analyzed (Participants) | 1
  Participant 2: 15 min post-dose (T7 liverP) | 0.01218
  Participant 2: 15 min post-dose (T8 liverR): number analyzed (Participants) | 1
  Participant 2: 15 min post-dose (T8 liverR) | 0.01079
  Participant 2: 1 hour post-dose (T1 lungL): number analyzed (Participants) | 1
  Participant 2: 1 hour post-dose (T1 lungL) | 0.00455
  Participant 2: 1 hour post-dose (T2 lungR): number analyzed (Participants) | 1
  Participant 2: 1 hour post-dose (T2 lungR) | 0.00463
  Participant 2: 1 hour post-dose (T3 liverL): number analyzed (Participants) | 1
  Participant 2: 1 hour post-dose (T3 liverL) | 0.01800
  Participant 2: 1 hour post-dose (T4 liverR1): number analyzed (Participants) | 1
  Participant 2: 1 hour post-dose (T4 liverR1) | 0.01400
  Participant 2: 1 hour post-dose (T5 liverR2): number analyzed (Participants) | 1
  Participant 2: 1 hour post-dose (T5 liverR2) | 0.01928
  Participant 2: 1 hour post-dose (T6 sacrumL): number analyzed (Participants) | 1
  Participant 2: 1 hour post-dose (T6 sacrumL) | 0.00289
  Participant 2: 1 hour post-dose (T7 liverP): number analyzed (Participants) | 1
  Participant 2: 1 hour post-dose (T7 liverP) | 0.01180
  Participant 2: 1 hour post-dose (T8 liverR): number analyzed (Participants) | 1
  Participant 2: 1 hour post-dose (T8 liverR) | 0.00961
  Participant 2: 2 hours post-dose (T1 lungL): number analyzed (Participants) | 1
  Participant 2: 2 hours post-dose (T1 lungL) | 0.00481
  Participant 2: 2 hours post-dose (T2 lungR): number analyzed (Participants) | 1
  Participant 2: 2 hours post-dose (T2 lungR) | 0.00377
  Participant 2: 2 hours post-dose (T3 liverL): number analyzed (Participants) | 1
  Participant 2: 2 hours post-dose (T3 liverL) | 0.00984
  Participant 2: 2 hours post-dose (T4 liverR1): number analyzed (Participants) | 1
  Participant 2: 2 hours post-dose (T4 liverR1) | 0.01527
  Participant 2: 2 hours post-dose (T5 liverR2): number analyzed (Participants) | 1
  Participant 2: 2 hours post-dose (T5 liverR2) | 0.02197
  Participant 2: 2 hours post-dose (T6 sacrumL): number analyzed (Participants) | 1
  Participant 2: 2 hours post-dose (T6 sacrumL) | 0.00254
  Participant 2: 2 hours post-dose (T7 liverP): number analyzed (Participants) | 1
  Participant 2: 2 hours post-dose (T7 liverP) | 0.01242
  Participant 2: 2 hours post-dose (T8 liverR): number analyzed (Participants) | 1
  Participant 2: 2 hours post-dose (T8 liverR) | 0.01088
  Participant 2: 4 hours post-dose (T1 lungL): number analyzed (Participants) | 1
  Participant 2: 4 hours post-dose (T1 lungL) | 0.00385
  articipant 2: 4 hours post-dose (T2 lungR): number analyzed (Participants) | 1
  articipant 2: 4 hours post-dose (T2 lungR) | 0.00248
  Participant 2: 4 hours post-dose (T3 liverL): number analyzed (Participants) | 1
  Participant 2: 4 hours post-dose (T3 liverL) | 0.01782
  Participant 2: 4 hours post-dose (T4 liverR1): number analyzed (Participants) | 1
  Participant 2: 4 hours post-dose (T4 liverR1) | 0.01164
  Participant 2: 4 hours post-dose (T5 liverR2): number analyzed (Participants) | 1
  Participant 2: 4 hours post-dose (T5 liverR2) | 0.02119
  Participant 2: 4 hours post-dose (T6 sacrumL): number analyzed (Participants) | 1
  Participant 2: 4 hours post-dose (T6 sacrumL) | 0.00188
  Participant 2: 4 hours post-dose (T7 liverP): number analyzed (Participants) | 1
  Participant 2: 4 hours post-dose (T7 liverP) | 0.01082
  Participant 2: 4 hours post-dose (T8 liverR): number analyzed (Participants) | 1
  Participant 2: 4 hours post-dose (T8 liverR) | 0.01012

8. Primary Outcome: Dosimetry Group: Evaluation of Percentage of Injected Dose Reaching the Target (TACs) in Organs
Description: For patients included in the dosimetry group, the percentage of injected dose per gram of tissue (%ID/g) reaching source organs was to be calculated using the acquired PET images at each time point. The resulting TACs were to be summarized descriptively.
Time Frame: [68Ga]-NeoBOMB1 PET imaging acquired at Day 1 (0.15, 1.00, 2.00 and 4.00 hours)
Population: as for outcome 7
Measure: Number; unit: %ID/g
Arm/Group | Breast
Number analyzed (Participants) | 2
%ID/g
  Participant 1: 15 min post-dose (Bladder): number analyzed (Participants) | 1
  Participant 1: 15 min post-dose (Bladder) | 0.03132
  Participant 1: 15 min post-dose (Heart): number analyzed (Participants) | 1
  Participant 1: 15 min post-dose (Heart) | 0.00600
  Participant 1: 15 min post-dose (Kidney): number analyzed (Participants) | 1
  Participant 1: 15 min post-dose (Kidney) | 0.00688
  Participant 1: 15 min post-dose (Liver): number analyzed (Participants) | 1
  Participant 1: 15 min post-dose (Liver) | 0.00794
  Participant 1: 15 min post-dose (Lung): number analyzed (Participants) | 1
  Participant 1: 15 min post-dose (Lung) | 0.00218
  Participant 1: 15 min post-dose (Marrow): number analyzed (Participants) | 1
  Participant 1: 15 min post-dose (Marrow) | 0.00331
  Participant 1: 15 min post-dose (Pancreas): number analyzed (Participants) | 1
  Participant 1: 15 min post-dose (Pancreas) | 0.04711
  Participant 1: 15 min post-dose (Spleen): number analyzed (Participants) | 1
  Participant 1: 15 min post-dose (Spleen) | 0.00409
  Participant 1: 1 hour post-dose (Bladder): number analyzed (Participants) | 1
  Participant 1: 1 hour post-dose (Bladder) | 0.04259
  Participant 1: 1 hour post-dose (Heart): number analyzed (Participants) | 1
  Participant 1: 1 hour post-dose (Heart) | 0.00241
  Participant 1: 1 hour post-dose (Kidney): number analyzed (Participants) | 1
  Participant 1: 1 hour post-dose (Kidney) | 0.00577
  Participant 1: 1 hour post-dose (Liver): number analyzed (Participants) | 1
  Participant 1: 1 hour post-dose (Liver) | 0.00296
  Participant 1: 1 hour post-dose (Lung): number analyzed (Participants) | 1
  Participant 1: 1 hour post-dose (Lung) | 0.00095
  Participant 1: 1 hour post-dose (Marrow): number analyzed (Participants) | 1
  Participant 1: 1 hour post-dose (Marrow) | 0.00116
  Participant 1: 1 hour post-dose (Pancreas): number analyzed (Participants) | 1
  Participant 1: 1 hour post-dose (Pancreas) | 0.04836
  Participant 1: 1 hour post-dose (Spleen): number analyzed (Participants) | 1
  Participant 1: 1 hour post-dose (Spleen) | 0.00211
  Participant 1: 2 hours post-dose (Bladder): number analyzed (Participants) | 1
  Participant 1: 2 hours post-dose (Bladder) | 0.02141
  Participant 1: 2 hours post-dose (Heart): number analyzed (Participants) | 1
  Participant 1: 2 hours post-dose (Heart) | 0.00163
  Participant 1: 2 hours post-dose (Kidney): number analyzed (Participants) | 1
  Participant 1: 2 hours post-dose (Kidney) | 0.00239
  Participant 1: 2 hours post-dose (Liver): number analyzed (Participants) | 1
  Participant 1: 2 hours post-dose (Liver) | 0.00197
  Participant 1: 2 hours post-dose (Lung): number analyzed (Participants) | 1
  Participant 1: 2 hours post-dose (Lung) | 0.00068
  Participant 1: 2 hours post-dose (Marrow): number analyzed (Participants) | 1
  Participant 1: 2 hours post-dose (Marrow) | 0.00092
  Participant 1: 2 hours post-dose (Pancreas): number analyzed (Participants) | 1
  Participant 1: 2 hours post-dose (Pancreas) | 0.05445
  Participant 1: 2 hours post-dose (Spleen): number analyzed (Participants) | 1
  Participant 1: 2 hours post-dose (Spleen) | 0.00141
  Participant 1: 4 hours post-dose (Bladder): number analyzed (Participants) | 1
  Participant 1: 4 hours post-dose (Bladder) | 0.01790
  Participant 1: 4 hours post-dose (Heart): number analyzed (Participants) | 1
  Participant 1: 4 hours post-dose (Heart) | 0.00130
  Participant 1: 4 hours post-dose (Kidney): number analyzed (Participants) | 1
  Participant 1: 4 hours post-dose (Kidney) | 0.00149
  Participant 1: 4 hours post-dose (Liver): number analyzed (Participants) | 1
  Participant 1: 4 hours post-dose (Liver) | 0.00162
  Participant 1: 4 hours post-dose (Lung): number analyzed (Participants) | 1
  Participant 1: 4 hours post-dose (Lung) | 0.00062
  Participant 1: 4 hours post-dose (Marrow): number analyzed (Participants) | 1
  Participant 1: 4 hours post-dose (Marrow) | 0.00035
  Participant 1: 4 hours post-dose (Pancreas): number analyzed (Participants) | 1
  Participant 1: 4 hours post-dose (Pancreas) | 0.06280
  Participant 1: 4 hours post-dose (Spleen): number analyzed (Participants) | 1
  Participant 1: 4 hours post-dose (Spleen) | 0.00120
  Participant 2: 15 min post-dose (Bladder): number analyzed (Participants) | 1
  Participant 2: 15 min post-dose (Bladder) | 0.02682
  Participant 2: 15 min post-dose (Heart): number analyzed (Participants) | 1
  Participant 2: 15 min post-dose (Heart) | 0.00340
  Participant 2: 15 min post-dose (Kidney): number analyzed (Participants) | 1
  Participant 2: 15 min post-dose (Kidney) | 0.00480
  Participant 2: 15 min post-dose (Liver): number analyzed (Participants) | 1
  Participant 2: 15 min post-dose (Liver) | 0.00866
  Participant 2: 15 min post-dose (Lung): number analyzed (Participants) | 1
  Participant 2: 15 min post-dose (Lung) | 0.00124
  Participant 2: 15 min post-dose (Marrow): number analyzed (Participants) | 1
  Participant 2: 15 min post-dose (Marrow) | 0.00186
  Participant 2: 15 min post-dose (Pancreas): number analyzed (Participants) | 1
  Participant 2: 15 min post-dose (Pancreas) | 0.02146
  Participant 2: 15 min post-dose (Spleen): number analyzed (Participants) | 1
  Participant 2: 15 min post-dose (Spleen) | 0.00338
  Participant 2: 1 hour post-dose (Bladder): number analyzed (Participants) | 1
  Participant 2: 1 hour post-dose (Bladder) | 0.06480
  Participant 2: 1 hour post-dose (Heart): number analyzed (Participants) | 1
  Participant 2: 1 hour post-dose (Heart) | 0.00207
  Participant 2: 1 hour post-dose (Kidney): number analyzed (Participants) | 1
  Participant 2: 1 hour post-dose (Kidney) | 0.00380
  Participant 2: 1 hour post-dose (Liver): number analyzed (Participants) | 1
  Participant 2: 1 hour post-dose (Liver) | 0.00564
  Participant 2: 1 hour post-dose (Lung): number analyzed (Participants) | 1
  Participant 2: 1 hour post-dose (Lung) | 0.00088
  Participant 2: 1 hour post-dose (Marrow): number analyzed (Participants) | 1
  Participant 2: 1 hour post-dose (Marrow) | 0.00136
  Participant 2: 1 hour post-dose (Pancreas): number analyzed (Participants) | 1
  Participant 2: 1 hour post-dose (Pancreas) | 0.02909
  Participant 2: 1 hour post-dose (Spleen): number analyzed (Participants) | 1
  Participant 2: 1 hour post-dose (Spleen) | 0.00256
  Participant 2: 2 hours post-dose (Bladder): number analyzed (Participants) | 1
  Participant 2: 2 hours post-dose (Bladder) | 0.04055
  Participant 2: 2 hours post-dose (Heart): number analyzed (Participants) | 1
  Participant 2: 2 hours post-dose (Heart) | 0.00142
  Participant 2: 2 hours post-dose (Kidney): number analyzed (Participants) | 1
  Participant 2: 2 hours post-dose (Kidney) | 0.00505
  Participant 2: 2 hours post-dose (Liver): number analyzed (Participants) | 1
  Participant 2: 2 hours post-dose (Liver) | 0.00428
  Participant 2: 2 hours post-dose (Lung): number analyzed (Participants) | 1
  Participant 2: 2 hours post-dose (Lung) | 0.00059
  Participant 2: 2 hours post-dose (Marrow): number analyzed (Participants) | 1
  Participant 2: 2 hours post-dose (Marrow) | 0.00100
  Participant 2: 2 hours post-dose (Pancreas): number analyzed (Participants) | 1
  Participant 2: 2 hours post-dose (Pancreas) | 0.03450
  Participant 2: 2 hours post-dose (Spleen): number analyzed (Participants) | 1
  Participant 2: 2 hours post-dose (Spleen) | 0.00191
  Participant 2: 4 hours post-dose (Bladder): number analyzed (Participants) | 1
  Participant 2: 4 hours post-dose (Bladder) | 0.11045
  Participant 2: 4 hours post-dose (Heart): number analyzed (Participants) | 1
  Participant 2: 4 hours post-dose (Heart) | 0.00093
  Participant 2: 4 hours post-dose (Kidney): number analyzed (Participants) | 1
  Participant 2: 4 hours post-dose (Kidney) | 0.00278
  Participant 2: 4 hours post-dose (Liver): number analyzed (Participants) | 1
  Participant 2: 4 hours post-dose (Liver) | 0.00317
  Participant 2: 4 hours post-dose (Lung): number analyzed (Participants) | 1
  Participant 2: 4 hours post-dose (Lung) | 0.00039
  Participant 2: 4 hours post-dose (Marrow): number analyzed (Participants) | 1
  Participant 2: 4 hours post-dose (Marrow) | 0.00072
  Participant 2: 4 hours post-dose (Pancreas): number analyzed (Participants) | 1
  Participant 2: 4 hours post-dose (Pancreas) | 0.03745
  Participant 2: 4 hours post-dose (Spleen): number analyzed (Participants) | 1
  Participant 2: 4 hours post-dose (Spleen) | 0.00145

9. Secondary Outcome: Treatment Emergent Adverse Events Profile
Description: Treatment-emergent adverse events (TEAEs) were collected from first dosing (single administration, Day 1) up to last follow-up visit or until the event has resolved to baseline grade or better or the event was assessed stable by the investigator or the patient was lost to follow-up or withdrew consent. The distribution of adverse events was done via the analysis of frequencies for treatment emergent Adverse Event (TEAEs), Grade 3/4/5 TEAEs, Serious Adverse Event TEAEs, Interruption of [68Ga]-NeoBOMB1 Due to Any TEAEs and Deaths due to AEs, through the monitoring of relevant clinical and laboratory safety parameters. Only descriptive analysis performed.
Time Frame: From first dosing (single administration, Day 1) up to last follow-up visit or until the event has resolved to baseline grade or better or the event was assessed stable by the investigator or the patient was lost to follow-up or withdrew consent.
Population: Full Analysis Set (FAS)
Measure: Count of Participants; unit: Participants
Arm/Group | Breast | Prostate | Colorectal | Non-Small Cell Lung Cancer (NSCLC) | Small-Cell Lung Cancer (SCLC)
Number analyzed (Participants) | 5 | 5 | 5 | 3 | 1
Participants
  Treatment-Emergent Adverse Events (TEAEs) | 0 | 1 | 3 | 3 | 1
  IMP-Related TEAEs | 0 | 0 | 0 | 0 | 0
  Grade 3/4/5 TEAEs | 0 | 0 | 0 | 0 | 1
  IMP-Related Grade 3/4/5 TEAEs | 0 | 0 | 0 | 0 | 0
  Serious TEAEs | 0 | 0 | 0 | 0 | 1
  IMP-Related Serious TEAEs | 0 | 0 | 0 | 0 | 0
  TEAEs Interruption of [68Ga]-NeoBOMB1 | 0 | 0 | 0 | 0 | 0
  IMP-Related TEAEs Interruption of [68Ga]-NeoBOMB1 | 0 | 0 | 0 | 0 | 0
  Deaths Due to AEs | 0 | 0 | 0 | 0 | 0

10. Secondary Outcome: Number of Lesions Detected by Conventional Imaging
Description: The preliminary targeting properties of [68Ga]-NeoBOMB1 were to be assessed by summarizing the number of lesions identified by Positron Emission Tomography (PET) overall and split by GRPR positive and negative patients, as well as by tumor type. The number of lesions identified by aforementioned PET imaging were to be compared with the number of lesions identified by the comparable conventional imaging. Only descriptive analysis performed.
Time Frame: Conventional imaging collected within 3 months prior to study entry up to [68Ga]-NeoBOMB1 PET imaging acquired at Day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Lesion
Arm/Group | Breast | Prostate | Colorectal | Non-Small Cell Lung Cancer (NSCLC) | Small-Cell Lung Cancer (SCLC)
Number analyzed (Participants) | 5 | 5 | 5 | 3 | 1
Lesion | 18.4 (15.81) | 13.8 (21.51) | 12.2 (9.86) | 10.0 (7.55) | 2.0 (NA) — Only one participant analyzed

11. Secondary Outcome: Number of Participants With Lesions Detected by Conventional Imaging Per Location
Description: The preliminary targeting properties of [68Ga]-NeoBOMB1 were to be assessed by summarizing the location of lesions identified by PET overall and split by GRPR positive and negative patients, as well as by tumor type. The location of lesions identified by aforementioned PET imaging were to be compared with the location of lesions identified by the comparable conventional imaging. Only descriptive analysis performed.
Time Frame: Conventional imaging collected within 3 months prior to study entry up to [68Ga]-NeoBOMB1 PET imaging acquired at Day 1
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Breast | Prostate | Colorectal | Non-Small Cell Lung Cancer (NSCLC) | Small-Cell Lung Cancer (SCLC)
Number analyzed (Participants) | 5 | 5 | 5 | 3 | 1
Participants
  Overall | 5 | 5 | 5 | 3 | 1
  Nodal | 4 | 1 | 2 | 3 | 1
  Skeletal | 4 | 2 | 0 | 0 | 0
  Skin/Superficial | 2 | 0 | 1 | 0 | 0
  Soft Tissue/Visceral | 4 | 4 | 5 | 3 | 1

12. Secondary Outcome: Lesion-level Analyses of Diagnostics by [68Ga]-NeoBOMB1 Compared With Conventional Imaging
Description: At lesion level, overall, positive, and negative agreement of [68Ga]-NeoBOMB1 were to be calculated based on the aforementioned tabulations as follows:
  * Overall agreement = 100% x (Double positive + Double negative) / total number of lesions identified by either imaging proceduresg
  * Positive agreement = 100% x Double positive / (Double positive + Comparator single positive)
  * Negative agreement = 100% x Double negative / (Double negative + Comparator single negative).
Time Frame: Conventional imaging collected within 3 months prior to study entry up to [68Ga]-NeoBOMB1 PET imaging acquired at Day 1
Population: Full Analysis Set (FAS).
Measure: Number (95% Confidence Interval); unit: Percent agreement
Arm/Group | Breast | Prostate | Colorectal | Non-Small Cell Lung Cancer (NSCLC) | Small-Cell Lung Cancer (SCLC)
Number analyzed (Participants) | 5 | 5 | 5 | 3 | 1
Percent agreement
  Overall (Positive Agreement) | 52.2 [41.5 to 62.7] | 14.5 [7.2 to 25.0] | 29.5 [18.5 to 42.6] | 33.3 [17.3 to 52.8] | 50.0 [1.3 to 98.7]
  Overall (Overall Agreement) | 37.2 [28.9 to 46.2] | 14.3 [7.1 to 24.7] | 29.5 [18.5 to 42.6] | 33.3 [17.3 to 52.8] | 50.0 [1.3 to 98.7]
  Nodal (Positive Agreement) | 64.3 [35.1 to 87.2] | 0.0 [0.0 to 30.8] | 66.7 [9.4 to 99.2] | 26.9 [11.6 to 47.8] | 0.0 [0.0 to 97.5]
  Nodal (Overall agreement) | 64.3 [35.1 to 87.2] | 0.0 [0.0 to 28.5] | 66.7 [9.4 to 99.2] | 26.9 [11.6 to 47.8] | 0.0 [0.0 to 97.5]
  Skeletal (Positive Agreement): number analyzed (Participants) | 5 | 5 | 0 | 0 | 0
  Skeletal (Positive Agreement) | 22.9 [12.0 to 37.3] | 11.1 [4.2 to 22.6] |  |  |
  Skeletal (Overall agreement): number analyzed (Participants) | 5 | 5 | 0 | 0 | 0
  Skeletal (Overall agreement) | 18.3 [9.5 to 30.4] | 11.1 [4.2 to 22.6] |  |  |
  Skin/Superficial (Positive Agreement): number analyzed (Participants) | 5 | 0 | 5 | 0 | 0
  Skin/Superficial (Positive Agreement) | 100.0 [15.8 to 100.0] |  | 0.0 [0.0 to 97.5] |  |
  Skin/Superficial (Overall agreement): number analyzed (Participants) | 5 | 0 | 5 | 0 | 0
  Skin/Superficial (Overall agreement) | 100.0 [15.8 to 100.0] |  | 0.0 [0.0 to 97.5] |  |
  Soft Tissue/Visceral (Positive Agreement) | 92.9 [76.5 to 99.1] | 80.0 [28.4 to 99.5] | 28.1 [17.0 to 41.5] | 75.0 [19.4 to 99.4] | 100.0 [2.5 to 100.0]
  Soft Tissue/Visceral (Overall agreement) | 49.1 [35.1 to 63.2] | 80.0 [28.4 to 99.5] | 28.1 [17.0 to 41.5] | 75.0 [19.4 to 99.4] | 100.0 [2.5 to 100.0]

13. Secondary Outcome: Patient-level Analyses of Diagnostics by [68Ga]-NeoBOMB1 Compared With Conventional Imaging
Description: At patient level, positive agreement was defined as the proportion of subjects with at least one lesion detected by conventional imaging in the specified location that also have at least one lesion detected by [68Ga]-NeoBOMB1. Overall agreement was defined as the proportion of subjects with at least one lesion detected in either imaging in the specified location that also have at least one lesion detected by [68Ga]-NeoBOMB1.
Time Frame: Conventional imaging collected within 3 months prior to study entry up to [68Ga]-NeoBOMB1 PET imaging acquired at Day 1
Population: Full Analysis Set (FAS).
Measure: Number (95% Confidence Interval); unit: Percent agreement
Arm/Group | Breast | Prostate | Colorectal | Non-Small Cell Lung Cancer (NSCLC) | Small-Cell Lung Cancer (SCLC)
Number analyzed (Participants) | 5 | 5 | 5 | 3 | 1
Percent agreement
  Overall (Positive Agreement) | 100.0 [47.8 to 100.0] | 100.0 [47.8 to 100.0] | 60.0 [14.7 to 94.7] | 100.0 [29.2 to 100.0] | 100.0 [2.5 to 100.0]
  Overall (Overall Agreement) | 100.0 [47.8 to 100.0] | 100.0 [47.8 to 100.0] | 60.0 [14.7 to 94.7] | 100.0 [29.2 to 100.0] | 100.0 [2.5 to 100.0]
  Nodal (Positive Agreement) | 50.0 [6.8 to 93.2] | 0.0 [0.0 to 97.5] | 100.0 [15.8 to 100.0] | 100.0 [29.2 to 100.0] | 0.0 [0.0 to 97.5]
  Nodal (Overall agreement) | 50.0 [6.8 to 93.2] | 0.0 [0.0 to 84.2] | 100.0 [15.8 to 100.0] | 100.0 [29.2 to 100.0] | 0.0 [0.0 to 97.5]
  Skeletal (Positive Agreement): number analyzed (Participants) | 5 | 5 | 0 | 0 | 0
  Skeletal (Positive Agreement) | 100.0 [39.8 to 100.0] | 100.0 [15.8 to 100.0] |  |  |
  Skeletal (Overall agreement): number analyzed (Participants) | 5 | 5 | 0 | 0 | 0
  Skeletal (Overall agreement) | 100.0 [39.8 to 100.0] | 100.0 [15.8 to 100.0] |  |  |
  Skin/Superficial (Positive Agreement): number analyzed (Participants) | 5 | 0 | 5 | 0 | 0
  Skin/Superficial (Positive Agreement) | 100.0 [15.8 to 100.0] |  | 0.0 [0.0 to 97.5] |  |
  Skin/Superficial (Overall agreement): number analyzed (Participants) | 5 | 0 | 5 | 0 | 0
  Skin/Superficial (Overall agreement) | 100.0 [15.8 to 100.0] |  | 0.0 [0.0 to 97.5] |  |
  Soft Tissue/Visceral (Positive Agreement) | 100.0 [39.8 to 100.0] | 100.0 [39.8 to 100.0] | 40.0 [5.3 to 85.3] | 100.0 [29.2 to 100.0] | 100.0 [2.5 to 100.0]
  Soft Tissue/Visceral (Overall agreement) | 100.0 [39.8 to 100.0] | 100.0 [39.8 to 100.0] | 40.0 [5.3 to 85.3] | 100.0 [29.2 to 100.0] | 100.0 [2.5 to 100.0]

14. Secondary Outcome: Organ-level Analyses of Diagnostics by [68Ga]-NeoBOMB1 Compared to Histological Evidence
Description: The diagnostic performance of [68Ga]-NeoBOMB1 to GRPR overexpressing malignancies (lesions) was to be compared with cytology and/or histopathology findings from archival and/or recent biopsy specimens.
  Since the biopsy was performed on 1 lesion (collected either in primary or in metastatic tumors), a direct link may not be possible in case of multiple lesions per organ identified on [68Ga]-NeoBOMB1-PET. In this event, the determination of positive versus negative lesions on [68Ga]-NeoBOMB1-PET was done at organ level, i.e., if any lesion is positive in that organ, then the organ was to be considered positive. The sensitivity was to be calculated as follows: Sensitivity = 100% x True positive / (True positive + False negative).
Time Frame: Biopsy specimen collected within 6 months prior to study entry up to [68Ga]-NeoBOMB1 PET imaging acquired at Day 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percent agreement
Arm/Group | Breast | Prostate | Colorectal | Non-Small Cell Lung Cancer (NSCLC) | Small-Cell Lung Cancer (SCLC)
Number analyzed (Participants) | 5 | 5 | 5 | 3 | 1
Percent agreement | 80.0 [28.4 to 99.5] | 100.0 [47.8 to 100.0] | 20.0 [0.5 to 71.6] | 100.0 [29.2 to 100.0] | 0.0 [0.0 to 97.5]

15. Secondary Outcome: Dosimetry Group: Absorbed Dose in Target Organs
Description: The absorbed dose in target organs and the effective radiation dose were to be summarized with descriptive statistics. Lesion number were assigned by dosimetry expert.
Time Frame: [68Ga]-NeoBOMB1 PET imaging acquired at Day 1
Population: as for outcome 7
Measure: Number; unit: mGy/MBq
Arm/Group | Breast
Number analyzed (Participants) | 2
mGy/MBq
  Participant 1-Alveolar interstital (Lungs): number analyzed (Participants) | 1
  Participant 1-Alveolar interstital (Lungs) | 0.0359
  Participant 1-Bone Marrow: number analyzed (Participants) | 1
  Participant 1-Bone Marrow | 0.0118
  Participant 1-Heart: number analyzed (Participants) | 1
  Participant 1-Heart | 0.0361
  Participant 1-Kidneys: number analyzed (Participants) | 1
  Participant 1-Kidneys | 0.0467
  Participant 1-Liver: number analyzed (Participants) | 1
  Participant 1-Liver | 0.0670
  Participant 1-Pancreas: number analyzed (Participants) | 1
  Participant 1-Pancreas | 0.3620
  Participant 1-Spleen: number analyzed (Participants) | 1
  Participant 1-Spleen | 0.0221
  Participant 1-Urinary bladder wall: number analyzed (Participants) | 1
  Participant 1-Urinary bladder wall | 0.0683
  Participant 2-Alveolar interstital (Lungs): number analyzed (Participants) | 1
  Participant 2-Alveolar interstital (Lungs) | 0.0241
  Participant 2-Bone Marrow: number analyzed (Participants) | 1
  Participant 2-Bone Marrow | 0.0064
  Participant 2-Heart: number analyzed (Participants) | 1
  Participant 2-Heart | 0.0158
  Participant 2-Kidneys: number analyzed (Participants) | 1
  Participant 2-Kidneys | 0.0339
  Participant 2-Liver: number analyzed (Participants) | 1
  Participant 2-Liver | 0.0450
  Participant 2-Pancreas: number analyzed (Participants) | 1
  Participant 2-Pancreas | 0.2270
  Participant 2-Spleen: number analyzed (Participants) | 1
  Participant 2-Spleen | 0.0189
  Participant 2-Urinary bladder wall: number analyzed (Participants) | 1
  Participant 2-Urinary bladder wall | 0.1010

16. Secondary Outcome: Dosimetry Group: Effective Whole-body Dose
Description: The effective radiation dose was to be summarized with descriptive statistics.
Time Frame: [68Ga]-NeoBOMB1 PET imaging acquired at Day 1
Population: as for outcome 7
Measure: Number; unit: mSv/MBq
Arm/Group | Breast
Number analyzed (Participants) | 2
mSv/MBq
  Participant 1: number analyzed (Participants) | 1
  Participant 1 | 0.0203
  Participant 2: number analyzed (Participants) | 1
  Participant 2 | 0.0151

17. Secondary Outcome: Dosimetry Group: Half-life of [68Ga]-NeoBOMB1 in Blood (T^1/2)
Description: Venous whole blood samples were collected for activity-based pharmacokinetics characterization in the dosimetry group. The half-lives of distribution (T^1/2 alpha) and elimination phases (T^1/2 beta) were to be listed and summarized using descriptive statistics.
Time Frame: [68Ga]-NeoBOMB1 PET imaging acquired at Day 1
Population: as for outcome 7
Measure: Number; unit: min
Arm/Group | Breast
Number analyzed (Participants) | 2
min
  Participant 1 - T^1/2 alpha: number analyzed (Participants) | 1
  Participant 1 - T^1/2 alpha | 7.39
  Participant 1 - T^1/2 beta: number analyzed (Participants) | 1
  Participant 1 - T^1/2 beta | 40.35
  Participant 2- T^1/2 alpha: number analyzed (Participants) | 1
  Participant 2- T^1/2 alpha | 1.73
  Participant 2- T^1/2 beta: number analyzed (Participants) | 1
  Participant 2- T^1/2 beta | 32.61

18. Secondary Outcome: Dosimetry Group: Time of Maximum Observed Drug Concentration Occurrence (Tmax)
Description: Venous whole blood samples were collected for activity-based pharmacokinetics characterization in the dosimetry group. Tmax was to be listed and summarized using descriptive statistics.
Time Frame: [68Ga]-NeoBOMB1 PET imaging acquired at Day 1
Population: as for outcome 7
Measure: Number; unit: min
Arm/Group | Breast
Number analyzed (Participants) | 2
min
  Participant 1: number analyzed (Participants) | 1
  Participant 1 | 5.78
  Participant 2: number analyzed (Participants) | 1
  Participant 2 | 5.73

19. Secondary Outcome: Dosimetry Group: Observed Maximum Plasma Concentration (Cmax)
Description: Venous whole blood samples were collected for activity-based pharmacokinetics characterization in the dosimetry group. Cmax was to be listed and summarized using descriptive statistics.
Time Frame: [68Ga]-NeoBOMB1 PET imaging acquired at Day 1
Population: as for outcome 7
Measure: Number; unit: kBq/cc
Arm/Group | Breast
Number analyzed (Participants) | 2
kBq/cc
  Participant 1: number analyzed (Participants) | 1
  Participant 1 | 15.95
  Participant 2: number analyzed (Participants) | 1
  Participant 2 | 31.31

20. Secondary Outcome: Dosimetry Group: Area Under the Plasma Concentration-time Curve From the Time 0 to the Last Observed Quantifiable Concentration (AUC(0-t))
Description: Venous whole blood samples were collected for activity-based pharmacokinetics characterization in the dosimetry group. AUC(0-t) was to be listed and summarized using descriptive statistics.
Time Frame: [68Ga]-NeoBOMB1 PET imaging acquired at Day 1
Population: as for outcome 7
Measure: Number; unit: MBq-s/cc
Arm/Group | Breast
Number analyzed (Participants) | 2
MBq-s/cc
  Participant 1: number analyzed (Participants) | 1
  Participant 1 | 40.67
  Participant 2: number analyzed (Participants) | 1
  Participant 2 | 44.85

21. Secondary Outcome: Dosimetry Group: AUC(0-t) Divided by the Dose Administered (AUC(0-t)/D)
Description: Venous whole blood samples were collected for activity-based pharmacokinetics characterization in the dosimetry group. AUC(0-t)/D was to be listed and summarized using descriptive statistics.
Time Frame: [68Ga]-NeoBOMB1 PET imaging acquired at Day 1
Population: as for outcome 7
Measure: Number; unit: s/cc
Arm/Group | Breast
Number analyzed (Participants) | 2
s/cc
  Participant 1: number analyzed (Participants) | 1
  Participant 1 | 0.2101
  Participant 2: number analyzed (Participants) | 1
  Participant 2 | 0.2301

22. Secondary Outcome: Dosimetry Group: Area Under the Concentration-time Curve From Time Zero (Pre-dose) Extrapolated to Infinite Time (AUCinf)
Description: Venous whole blood samples were collected for activity-based pharmacokinetics characterization in the dosimetry group. AUC(0-inf) was to be listed and summarized using descriptive statistics.
Time Frame: [68Ga]-NeoBOMB1 PET imaging acquired at Day 1
Population: as for outcome 7
Measure: Number; unit: MBq-s/cc
Arm/Group | Breast
Number analyzed (Participants) | 2
MBq-s/cc
  Participant 1 | 44.49
  Participant 2 | 70.21

23. Secondary Outcome: Dosimetry Group: Total Systemic Clearance for Intravenous Administration (CL)
Description: Venous whole blood samples were collected for activity-based pharmacokinetics characterization in the dosimetry group. CL was to be listed and summarized using descriptive statistics.
Time Frame: [68Ga]-NeoBOMB1 PET imaging acquired at Day 1
Population: as for outcome 7
Measure: Number; unit: cc/s
Arm/Group | Breast
Number analyzed (Participants) | 2
cc/s
  Participant 1: number analyzed (Participants) | 1
  Participant 1 | 43.50
  Participant 2: number analyzed (Participants) | 1
  Participant 2 | 2.78

24. Secondary Outcome: Dosimetry Group: Urinary Excretion of [68Ga]-NeoBOMB1 (Vd)
Description: Urine samples were collected for activity-based pharmacokinetics characterization in the dosimetry group. Vd was to be listed and summarized using descriptive statistics.
Time Frame: [68Ga]-NeoBOMB1 PET imaging acquired at Day 1
Population: Full Analysis Set (FAS). Dosimetry group targeted participants with Breast Cancer and Prostate Cancer, but only 2 participants from Breast Cancer arm enrolled in the Dosimetry Group. As the total volume of excreted urine was not recorded, no percentage of urinary excretion could be calculated.
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Breast
Number analyzed (Participants) | 2
L | NA (NA) — NA: total volume of excreted urine was not recorded. Thus, no % of urinary excretion could be calculated.

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected from informed consent signature through study completion (Day 14).
Description: Any sign or symptom that occurs after written informed consent provided. For TEAE from first dosing (single administration, Day 1) up to last follow-up visit or until the event has resolved to baseline grade or better or the event was assessed stable by the investigator or the patient was lost to follow-up or withdrew consent.
Arm/Group | Breast | Prostate | Colorectal | Non-Small Cell Lung Cancer (NSCLC) | Small-Cell Lung Cancer (SCLC)
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5 | 0/5 | 0/3 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5 | 0/5 | 0/3 | 1/1
Other Adverse Events (participants affected / at risk) | 0/5 | 1/5 | 3/5 | 3/3 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Breast (N=5) | Prostate (N=5) | Colorectal (N=5) | Non-Small Cell Lung Cancer (NSCLC) (N=3) | Small-Cell Lung Cancer (SCLC) (N=1)
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Breast (N=5) | Prostate (N=5) | Colorectal (N=5) | Non-Small Cell Lung Cancer (NSCLC) (N=3) | Small-Cell Lung Cancer (SCLC) (N=1)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Hyperfibrinogenaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 1
Hyperparathyroidism (Endocrine disorders) | 0 | 1 | 0 | 0 | 1
Post procedural constipation (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Blood cholinesterase decreased (Investigations) | 0 | 0 | 0 | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 1 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 1 | 0
Blood urea decreased (Investigations) | 0 | 0 | 0 | 0 | 1
C-reactive protein increased (Investigations) | 0 | 0 | 0 | 1 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 1 | 0 | 1
Hyperalbuminaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Hypochloraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Paralysis recurrent laryngeal nerve (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0 | 0

LIMITATIONS AND CAVEATS:
Recruitment was stopped before the target sample size was achieved..

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Statistical Analysis Plan (2019-06-11): https://cdn.clinicaltrials.gov/large-docs/53/NCT03724253/SAP_000.pdf
  • Study Protocol (2018-07-05): https://cdn.clinicaltrials.gov/large-docs/53/NCT03724253/Prot_001.pdf